CLINICAL TRIAL: NCT02596230
Title: Characterization of Patients Following Acute Venous Thromboembolism (VTE) and Safety and Effectiveness of Dabigatran Etexilate (DE) in the Treatment and Secondary Prevention of Acute Deep Vein Thrombosis (DVT) and Pulmonary Embolism (PE) in Comparison to Vitamin K Antagonist (VKA) in Routine Clinical Practice - RE-COVERY DVT/PE
Brief Title: RE-COVERY DVT/PE: Global Study on Treatment Secondary Prevention of Acute Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.188
Record Dates: First submitted 2015-10-28; First posted 2015-11-04 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Patients with acute VTE: Patients will be enrolled for cross sectional characterization of baseline characteristics
- Dabigatran: Patients treated with dabigatran for acute VTE will be followed for one year
- vitamin K antagonist: Patients treated with VKA for acute VTE will be followed for one year

SUMMARY:
RE-COVERY is a large, multi-national, multi-center observational study based on new data collection. The study will enroll and characterize patients within 30 days of being diagnosed with an acute DVT and/or PE. The study has two main objectives. Objective 1 will characterize the DVT / PE patient population. All patients with a DVT and/or PE will be enrolled for cross-sectional characterization of the VTE patient population. Objective 2 will compare the safety and effectiveness of dabigatran etexilate regimens for treatment of VTE in comparison to VKA regimens. Patients treated with dabigatran etexilate or VKA will be followed up for the occurrence of outcome events for up to one year.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent provided by the patient in accordance with local regulations
2. Diagnosis of an acute DVT and/or PE (For objective 1, assessment of patient for study participation should be done ideally within 14 days but not more than 6 months after diagnosis of the acute VTE. For Objective 2, patient assessment should occur ideally within 14 days but not more than 30 days from diagnosis)
3. Age >= 18 years
4. For Objective 2, the planned anticoagulation therapy should be for at least 3 months
5. For Objective 2, dabigatran and vitamin K antagonist patients should be available for follow-up data collection

Exclusion criteria:

1. Need for anticoagulation therapy for conditions other than venous thromboembolism (VTE)
2. Current participation in a clinical trial for VTE indication or current use of an unapproved drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute venous thromboembolism
Sampling Method: Non-Probability Sample
Enrollment: 7797 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (222):
- United States (19):
  - Cardiovascular Innovation and Research Center, Long Beach, California
  - Health and Life Research Institute, LLC, Miami, Florida
  - Med-Care Research, Miami, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Tampa General Hospital, Tampa, Florida
  - Ellipsis Group, Atlanta, Georgia
  - Wellstar Cardiovascular Medicine, Marietta, Georgia
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Vidant Multispecialty Clnc Kinston, Kinston, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Lycoming Internal Medicine, Inc, Jersey Shore, Pennsylvania
  - Research Associates of Jackson, Jackson, Tennessee
  - The University Of Texas at Houston, Houston, Texas
  - Cardiology Center of Houston, PA, Katy, Texas
  - Cardio Voyage, McKinney, Texas
  - Waukesha Heart Institute, Waukesha, Wisconsin
- Argentina (5):
  - Hospital Universitario Austral, Buenos Aires
  - Hospital Aleman, CABA
  - Hospital Italiano, CABA
  - ICBA, CABA
  - Clinica Juncal, Temperley
- Austria (3):
  - LKH Feldkirch, Feldkirch
  - LKH-Univ. Hospital Graz, Graz
  - Medical University of Innsbruck, Innsbruck
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - C.H.U. de Charleroi, Charleroi
  - H.-Hartziekenhuis, Lier
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (3):
  - Hospital Vera Cruz, Belo Horizonte
  - Faculdade de Ciencias Medicas da UNICAMP, Campinas
  - Hospital das Clinicas da Faculdade de Medicina - FMUSP, São Paulo
- Bulgaria (4):
  - UMHAT St. George, Plovdiv
  - National Heart Hospital, Sofia, Sofia
  - MHAT 'Tokuda Hospital Sofia', EAD, Sofia
  - Hospital Trakia Park, Stara Zagora
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital - Hamilton Health Sciences, Hamilton, Ontario
- SMOLAM, Santiago, Chile
- Colombia (6):
  - Fundacion Cardiomet CEQUIN, Armenia
  - Unidad de Investigaciones Clínicas, Cali
  - Centro de Investigaciones Clinicas S.A.S, Cali
  - Centro de Diagnostico Cardilogico, Cartagena
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
  - Promotora Medica Las Americas SA, Medellín
- Czechia (13):
  - Rehabilitacni nemocnice Beroun, Beroun
  - Diagangio s.r.o., Brno
  - University Hospital Brno, Brno
  - Nemocnice Milosrdnych bratri, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - CTC Hodonin s.r.o., Hodonín
  - MUDr. Ladislav Busak, Louny
  - MUDr. Stanislav Bulir, Mladá Boleslav
  - Nemocnice Náchod, Náchod
  - MUDr. Dalibor Musil, Olomouc
  - Fakultni nemocnice Plzen, Pilsen
  - Vseobecna fakultni nemocnice V Praze, Prague
  - Institute for Clinical and Experimental Medicine, Prague
- Egypt (5):
  - Dr. Ashraf ElGhandour Private Clinic, Alexandria
  - Private Clinic Dr. Mervat Mattar, Cairo
  - Private Clinic Mohamed Moussa, Cairo
  - Private Clinic - Dr. Shawky, Cairo
  - Private Clinic - Dr. Ahmed Hassouna, Kalyoub
- Germany (5):
  - Franziskus-Krankenhaus, Berlin, Berlin
  - Städtisches Klinikum Dresden, Dresden
  - Praxis für Gefäßmedizin, Görlitz
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Heidelberg, Heidelberg
- Greece (9):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - "Laiko" Hospital, 1st Vascular Surgery Clinic of UOA, Athens
  - Athens Hospital of Chest Diseases "Sotiria", Athens
  - Gen. Hosp. of Chest Diseases "Sotiria", 3rd Internal Med. Cl, Athens
  - University General Hospital Attikon, Athens
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - General Hospital of Athens "G. Gennimatas", Thessaloniki
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Hungary (9):
  - Dr. Kenessey Albert Kórház-Rendelõintézet, Balassagyarmat, Balassagyarmat
  - St. Istvan Hospital, Budapest, Budapest
  - Jahn Ferenc Del-Pest Hospital, Budapest
  - University Debrecen Hospital, Debrecen
  - Pest Megyei Flor Ferenc Hospital, Kistarcsa
  - Dorottya Kanizsai Hospital, Nagykanizsa
  - Pecsi Tudomanyegyetem, Pécs
  - Csongrad Country Dr Bugyi Istvan Hosp., Szentes
  - Jasz-Nagykun-Szolnok Megyei Hetenyi G. Korhaz-Rendelointezet, Szolnok
- Italy (16):
  - Clinica Villa dei Fiori, Acerra
  - Ospedale san Lazzaro, Alba
  - Policlinico di Bari, Bari
  - P.O. di Castelfranco Veneto, Castelfranco Veneto
  - Ospedale Civile degli Infermi, Faenza (RA)
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Spedali Riuniti di Livorno, Livorno
  - Ospedali Riuniti di Ancona, Macerata
  - SUN Seconda Università Napoli, Napoli
  - Ospedale Gaetano Bernabeo, Ortona (CH)
  - Osp. Civico e Benfratelli "M. Ascoli e G. Di Cristina", Palermo
  - Azienda Universitaria-Universita' La Sapienza, Roma
  - Univ. Cattolica del Sacro Cuore, Roma
  - Ospedale Civile, Sassari
  - A. O. Ospedale Circolo Fond. Macchi, Varese
  - A. O. Ospedale di Vimercate, Vimercate (Mi)
- Latvia (5):
  - Daugavpils Regional Hospital, Daugavpils
  - Liepaja Regional Hospital, Therapy Department, Liepāja
  - Riga East University Hospital, Riga
  - VSV Centrs, Stalte Private Practice, Talsi, Talsi
  - Gita Rancane Doctor Practice in Cardiology, Ventspils
- Lebanon (7):
  - Clemenceau Medical Center, Beirut
  - Rafik Hariri University Hospital, Beirut
  - American University of Beirut Medical Center, Beirut
  - Bellevue Medical Center, Beirut
  - Centre Hospitalier Universitaire Notre Dame de Secours, Byblos
  - Ain Wazein Hospital, El-Chouf
  - Hammoud Hospital University Medical Center, Saida
- Malaysia (2):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kota Bharu
  - University Malaya Medical Centre, Kuala Lumpur
- Mexico (4):
  - Clinica Vascular de Guadalajara, Guadalajara
  - Instituto Jalisciense de Metabolismo, SC, Guadalajara
  - Hospital_Angeles Centro Médicodel Potosí, San Luis Potosí City
  - Arke Estudios Clinicos SA de CV, Veracruz
- Netherlands (4):
  - OLVG, locatie Oosterpark, Amsterdam
  - Amphia Ziekenhuis, Breda
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Tweesteden Ziekenhuis, locatie Tilburg, Tilburg
- Palmerston North Hospital, Palmerston North, New Zealand
- Centro Medico Piura, Piura, Peru
- Philippines (3):
  - Makati Medical Center, Makati
  - Philippine General Hospital, Manila, Philippines
  - St. Luke's Medical Center, QC, Quezon City
- Poland (4):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 4, Bytom
  - Mazowiecki Szpital Specjalistyczny im. dr Jozefa Psarskiego, Ostrołęka
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
- Portugal (4):
  - Hospital Ponta Delgada, Ponta Delgada
  - Centro Hospitalar Universitário do Porto, EPE - Hospital de Santo António, Porto
  - Hospital CUF Porto, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Romania (3):
  - Private Practice Cardiology Dr. Pop Calin Florin, Baia Mare
  - Emergency University Hospital, Bucharest, Bucharest
  - Spitalul Clinic Municipal Cluj Napoca, Cluj-Napoca
- Russia (18):
  - Regional Clinical Hospital#3, Chelyabinsk
  - State Autonomous Institution of Health, Kemerovo
  - Hospital #15 named after O.M.Filatov, Moscow
  - Federal Research and Clinical Center of Special Medical Help, Moscow
  - City Clinical Hospital 1 (1-Gradskaya), Moscow
  - City Clinical Hospital n.a. V.V. Veresaev, Moscow
  - Novosibirsk Research Institute, Novosibirsk
  - Rostov Medical University, Rostov-on-Don
  - City Clinical Hospital No. 2, St. Petersburg, Saint Petersburg
  - St.Petersburg State Medical University n. a. II Mechnikov, Saint Petersburg
  - City Hospital Saint Elizaveta, Dept. Endocrinology, Saint Petersburg
  - Dorozghnaya hospital, Saint Petersburg
  - Clinical hospital of BGMU, Ufa
  - Clinical emergency hospital #15, Volgograd
  - Voronezh Regional Hospital N1, Voronezh
  - Yaroslavl Regional Clin. Hospital, Yaroslavl
  - Medical Center "Angioline", Yekaterinburg
  - LLC Medical Union New Hospital, Yekaterinburg
- King Fahad Medical City, Riyadh, Saudi Arabia
- Serbia (9):
  - Clinical Center of Serbia, Belgrade
  - Clinical Medical Center Zvezdara, Belgrade, Belgrade
  - Institute for Cardiovascular diseases Dedinje, Belgrade
  - General Hospital MediGroup, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade, Belgrade
  - Inst. for Pulm. Diseases of Vojvodine, Clinic f. Pulm. Oncol, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Centre Nis, Niš
  - General Hospital Valjevo, Valjevo
- Slovakia (5):
  - ALIAN s.r.o., Bardejov, Dzupinova, Maria, Bardejov
  - KARDIO-ANGIO, s.r.o., Levice
  - HeMart, s.r.o., Martin
  - ABE-AS, s.r.o., Nitra
  - MEDIVASA s.r.o., Outpatient Clinic, Zilina, Žilina
- Slovenia (4):
  - GH Celje, Celje
  - Univ. Clinic of Respiratory and Allergic Diseases, Golnik, Golnik
  - UCC Maribor, Maribor
  - Hospital Topolsica, Topolšica
- South Korea (10):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Thammasat University Hospital, Pathum Tani
- Turkey (Türkiye) (14):
  - Gazi University Medical Faculty, Ankara
  - Ankara Atatürk Training and Research Hospital, Ankara
  - Uludag University Medical Faculty, Bursa
  - Dicle University Medical Faculty, Diyarbakır
  - Dr. Ersin Arslan Public Hospital, Gaziantep
  - Suleyman Demirel University Medical Faculty, Isparta
  - Bakirköy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi Zuhura, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Izmir Tepecik Training and Research Hospital, Izmir
  - Ege University Medical Faculty, Izmir
  - Karaman Government Hospital, Karaman
  - Kayseri Training And Research Hospital, Kayseri
  - RTE University Medical Faculty, Rize
  - Ozel Uzmanlar Yalova Hospital, Yalova
- Thumbay Hospital, Dubai, United Arab Emirates
- United Kingdom (10):
  - Barnsley Hospital, Barnsley
  - North Hampshire Hospital, Basingstoke
  - Birmingham Heartlands Hospital, Birmingham
  - Queen's Hospital, Burton-on-Trent
  - University Hospital of North Durham, Durham
  - St Thomas' Hospital, London
  - Wythenshawe Hospital, Manchester
  - North Tyneside General Hospital, North Shields
  - Craigavon Area Hospital, Portadown
  - Salisbury District Hospital, Salisbury
- Vietnam (5):
  - Bach Mai hospital, Hanoi
  - 115 People Hospital, Ho Chi Minh City
  - Gia Dinh People Hospital, Ho Chi Minh City
  - Cho Ray Hospital, Ho Chi Minh City
  - University Medical Center of Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goldhaber SZ, Ageno W, Casella IB, Chee KH, Schellong S, Singer DE, Voccia I, Tang W, Schulman S. Safety and effectiveness of dabigatran in routine clinical practice: the RE-COVERY DVT/PE study. J Thromb Thrombolysis. 2022 Feb;53(2):399-409. doi: 10.1007/s11239-021-02463-x. Epub 2021 Aug 28. PMID 34453675
- [Derived] Ageno W, Casella IB, Chee KH, Schellong S, Schulman S, Singer DE, Desch M, Tang W, Voccia I, Zint K, Goldhaber SZ. Profile of patients diagnosed with acute venous thromboembolism in routine practice according to age and renal function: RE-COVERY DVT/PE study. J Thromb Thrombolysis. 2021 Apr;51(3):561-570. doi: 10.1007/s11239-020-02239-9. PMID 32851572
- [Derived] Goldhaber SZ, Ageno W, Casella IB, Chee KH, Schellong S, Singer DE, Desch M, Reilly PA, Donado E, Tang W, Voccia I, Schulman S. Profile of Patients Diagnosed With Acute Venous Thromboembolism in Routine Clinical Practice: The RE-COVERY DVT/PE Study. Am J Med. 2020 Aug;133(8):936-945. doi: 10.1016/j.amjmed.2020.03.036. Epub 2020 Apr 20. PMID 32325043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study characterizes patients following acute venous thromboembolism and assesses the safety and effectiveness of dabigatran etexilate in the treatment and secondary prevention of acute DVT and PE in comparison to vitamin K antagonist in routine clinical practice. This is a large multi-center observational study based on new data collection.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that they met all inclusion/exclusion criteria. The study enrolled and characterized all patients within 30 days after being diagnosed with an acute DVT and/or PE.
Groups:
- Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist: Participants diagnosed with an acute Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE) and treated with either Edoxaban, Rivaroxaban, Apixaban or other anticoagulation treatments. Participants analyzed for objective 1 only.
- Dabigatran Etexilate (1): Participants diagnosed with an acute Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE) and treated with Dabigatran etexilate. Participants analyzed for objective 1 or for objective 1 and 2.
- Dabigatran Etexilate (2): Participants diagnosed with an acute Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE) and treated with Dabigatran etexilate. New participants analyzed for objective 2 only.
- Vitamin K Antagonist (1): Participants diagnosed with an acute Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE) and treated with Vitamin K antagonist. Participants analyzed for objective 1 or for objective 1 and 2.
- Vitamin K Antagonist (2): Participants diagnosed with an acute Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE) and treated with Vitamin K antagonist. New participants analyzed for objective 2 only.
Period: Objective 1, One Visit During 14 Days
Arm/Group | Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist | Dabigatran Etexilate (1) | Dabigatran Etexilate (2) | Vitamin K Antagonist (1) | Vitamin K Antagonist (2)
Started | 3714 | 1006 | 0 | 1375 | 0
Completed | 3714 | 1006 | 0 | 1375 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Screening Period for Objective 2
Arm/Group | Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist | Dabigatran Etexilate (1) | Dabigatran Etexilate (2) | Vitamin K Antagonist (1) | Vitamin K Antagonist (2)
Started | 3714 | 1006 | 910 (Participants entering the study after the completion of objective 1.) | 1375 | 792 (Participants entering the study after the completion of objective 1.)
Completed | 0 | 778 | 910 | 529 | 792
Not Completed | 3714 | 228 | 0 | 846 | 0
Not completed — Participants not participating in obj 2 | 3714 | 228 | 0 | 846 | 0
Period: Objective 2, One Year
Arm/Group | Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist | Dabigatran Etexilate (1) | Dabigatran Etexilate (2) | Vitamin K Antagonist (1) | Vitamin K Antagonist (2)
Started | 0 | 778 | 910 | 529 | 792
Completed | 0 | 710 | 812 | 471 | 714
Not Completed | 0 | 68 | 98 | 58 | 78
Not completed — Lost to Follow-up | 0 | 41 | 41 | 32 | 46
Not completed — Withdrawal by Subject | 0 | 11 | 14 | 5 | 2
Not completed — Adverse drug reaction | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 12 | 41 | 21 | 30
Not completed — Other | 0 | 3 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Eligible: patients fulfilling all inclusion criteria and no exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist | Dabigatran Etexilate (1) | Dabigatran Etexilate (2) | Vitamin K Antagonist (1) | Vitamin K Antagonist (2) | Total
Number analyzed (Participants) | 3714 | 1006 | 910 | 1375 | 792 | 7797
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (17.2) | 58.3 (16.6) | 58.4 (16.6) | 61.3 (16.6) | 59.0 (16.6) | 60.9 (17.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1806 | 548 | 477 | 708 | 417 | 3956
  Female | 1907 | 458 | 433 | 667 | 375 | 3840
  Missing | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 2 | 7 | 14
  Asian | 420 | 149 | 147 | 96 | 124 | 936
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 0 | 0 | 0 | 4
  Black or African American | 111 | 2 | 7 | 71 | 18 | 209
  White | 2620 | 828 | 742 | 1152 | 600 | 5942
  More than one race | 5 | 6 | 11 | 7 | 42 | 71
  Unknown or Not Reported | 552 | 20 | 1 | 47 | 1 | 621

OUTCOME MEASURES:

1. Primary Outcome: Objective 1: Age
Description: Age in years of eligible patients collected for Objective 1 during baseline at the time of index event. Aim of Objective 1 was to characterize the Venous Thromboembolism (VTE) patient population including the initial acute event phase, i.e. all patients regardless of treatment. Patients who enrolled in Objective 1 and were treated with VKA or dabigatran were also eligible for Objective 2. The aim of objective 2 was to analyze the safety and effectiveness of dabigatran regimens in the treatment of DVT and PE over 1 year of follow-up in comparison to a VKA regimen.
  The arm presented in this endpoint was separated into three arms in the participant flow tables ("Not assigned to Dabigatran etexilate or Vitamin K antagonist","Dabigatran etexilate (1)" and "Vitamin K antagonist (1)") in order to distinguish patients participating in both objectives from patients only in objective 2.
Time Frame: Baseline collected within 14 days but not more than 6 months after diagnosis of acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE).
Population: All eligible patients with a DVT and/or PE (regardless of treatment) were enrolled for cross-sectional characterisation of the VTE patient population
Measure: Mean (Standard Deviation); unit: years
Groups:
- All Participants With a DVT and/or PE: All participants diagnosed with Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE).
Arm/Group | All Participants With a DVT and/or PE
Number analyzed (Participants) | 6095
years | 61.5 (17.0)

2. Primary Outcome: Objective 1: Sex
Description: Sex of eligible patients collected for Objective 1 during baseline at the time of index event. Aim of Objective 1 was to characterize the Venous Thromboembolism (VTE) patient population including the initial acute event phase, i.e. all patients regardless of treatment. Patients who enrolled in Objective 1 and were treated with VKA or dabigatran were also eligible for Objective 2. The aim of objective 2 was to analyze the safety and effectiveness of dabigatran regimens in the treatment of DVT and PE over 1 year of follow-up in comparison to a VKA regimen.
  The arm presented in this endpoint was separated into three arms in the participant flow tables ("Not assigned to Dabigatran etexilate or Vitamin K antagonist","Dabigatran etexilate (1)" and "Vitamin K antagonist (1)") in order to distinguish patients participating in both objectives from patients only in objective 2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With a DVT and/or PE
Number analyzed (Participants) | 6095
Participants
  Male: Participants | 3062
  Female: Participants | 3032
  Missing data: Participants | 1

3. Primary Outcome: Objective 1: Index Event
Description: Type of index event (e.g., DVT or PE or DVT and PE) diagnosed at the time of acute Venous Thromboembolism (VTE) event of eligible patients collected for Objective 1 during baseline at the time of index event. Aim of Objective 1 was to characterize the Venous Thromboembolism (VTE) patient population including the initial acute event phase, i.e. all patients regardless of treatment. Patients who enrolled in Objective 1 and were treated with VKA or dabigatran were also eligible for Objective 2. The aim of objective 2 was to analyze the safety and effectiveness of dabigatran regimens in the treatment of DVT and PE over 1 year of follow-up in comparison to a VKA regimen.
  The arm presented in this endpoint was separated into three arms in the participant flow tables ("Not assigned to Dabigatran etexilate or Vitamin K antagonist","Dabigatran etexilate (1)" and "Vitamin K antagonist (1)") in order to distinguish patients participating in both objectives from patients only in objective 2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With a DVT and/or PE
Number analyzed (Participants) | 6095
Participants
  DVT: Participants | 3644
  PE: Participants | 1588
  DVT and PE: Participants | 863

4. Primary Outcome: Objective 1: Anticoagulant Treatment
Description: Type of treatment received following acute Venous Thromboembolism (VTE) event of eligible patients collected for Objective 1 during baseline at the time of index event. Aim of Objective 1 was to characterize the Venous Thromboembolism (VTE) patient population including the initial acute event phase, i.e. all patients regardless of treatment. Patients who enrolled in Objective 1 and were treated with VKA or dabigatran were also eligible for Objective 2. The aim of objective 2 was to analyze the safety and effectiveness of dabigatran regimens in the treatment of DVT and PE over 1 year of follow-up in comparison to a VKA regimen.
  The arm presented in this endpoint was separated into three arms in the participant flow tables ("Not assigned to Dabigatran etexilate or Vitamin K antagonist","Dabigatran etexilate (1)" and "Vitamin K antagonist (1)") in order to distinguish patients participating in both objectives from patients only in objective 2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With a DVT and/or PE
Number analyzed (Participants) | 6095
Participants
  Dabigatran: Participants | 947
  vitamin K antagonist (VKA): Participants | 1388
  Edoxaban: Participants | 103
  Rivaroxaban: Participants | 1558
  Apixaban: Participants | 686
  Other: Participants | 1413

5. Primary Outcome: Objective 2: Incidence Rate of ISTH (International Society on Thrombosis and Haemostasis) Major Bleeding and CRNMB (Clinically Relevant Non Major Bleeding) Per 100 Patient-years (Pt-yrs)
Description: Incidence rate of ISTH (International Society on Thrombosis and Haemostasis) major bleeding and CRNMB (clinically relevant non major bleeding) per 100 patient-years (1/(100*patient-years)). Each patient in the two treatment groups was weighted proportionally to the probability of that patient being assigned to the opposite treatment group, conditional on relevant observed baseline variables. The propensity scores were estimated using the multivariable logistic regression model.
  For the restricted patient set, as a sensitivity analysis, the calculation of incidence rates and cumulative risks was performed without censoring at permanent discontinuation.
Time Frame: 12 months following acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE).
Population: Restricted set: The restricted population was composed of all eligible patients, which lay within the region of propensity score overlap and who took the prescribed treatment at least once.
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Groups:
- Dabigatran Etexilate: Participants diagnosed with an acute Deep Vein Thrombosis (DVT) irrespective of location and/or Pulmonary Embolism (PE) and treated with Dabigatran etexilate. This includes both participants who participated in objective 1 and 2 and new participants only participating in objective 2.
- Vitamin K Antagonist: Participants diagnosed with an acute DVT and/or PE and treated with Vitamin K antagonist. This includes both participants who participated in objective 1 and 2 and new participants only participating in objective 2.
Arm/Group | Dabigatran Etexilate | Vitamin K Antagonist
Number analyzed (Participants) | 1681 | 1288
events per 100 patient-years | 2.63 [1.79 to 3.73] | 4.42 [3.18 to 5.97]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Vitamin K Antagonist; Test type: Other; p = 0.188, Regression, Cox — One-side p-value; Cox-regression proportional hazards model including fixed effects for treatment; Hazard Ratio (HR) = 0.634, 95% CI 2-sided [0.322 to 1.249] — Hazard Ratio < 1 favors Dabigatran etexilate

6. Primary Outcome: Objective 2: Symptomatic Recurrent VTE (Venous Thromboembolism) Including VTE Related Mortality
Description: Incidence rate of Symptomatic Recurrent VTE (Venous Thromboembolism) including VTE related mortality per 100 patient-years (1/(100*patient-years)). Each patient in the two treatment groups was weighted proportionally to the probability of that patient being assigned to the opposite treatment group, conditional on relevant observed baseline variables. The propensity scores were estimated using the multivariable logistic regression model.
  For the restricted patient set, as a sensitivity analysis, the calculation of incidence rates and cumulative risks was performed without censoring at permanent discontinuation.
Time Frame: 12 months following acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE).
Population: Restricted set: The restricted population was composed of all eligible patients, which lay within the region of propensity score overlap. The propensity scores are estimated after the multiple imputation is performed based on eligible patients who took the prescribed treatment at least once.
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Dabigatran Etexilate | Vitamin K Antagonist
Number analyzed (Participants) | 1681 | 1288
events per 100 patient-years | 1.53 [0.91 to 2.42] | 2.01 [1.21 to 3.14]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Vitamin K Antagonist; Test type: Other; p = 0.606, Regression, Cox — One-side p-value; Cox-regression proportional hazards model including fixed effects for treatment; Hazard Ratio (HR) = 0.778, 95% CI 2-sided [0.300 to 2.017] — Hazard Ratio < 1 favors Dabigatran etexilate

7. Secondary Outcome: Objective 2: Incidence Rate of Recurrent DVT and/or PE
Description: Incidence rate of Recurrent Deep Vein Thrombosis (DVT) and/or Pulmonary Embolism (PE) per 100 patient-years (1/(100*patient-years)). Each patient in the two treatment groups was weighted proportionally to the probability of that patient being assigned to the opposite treatment group, conditional on relevant observed baseline variables. The propensity scores were estimated using the multivariable logistic regression model.
  For the restricted patient set, as a sensitivity analysis, the calculation of incidence rates and cumulative risks was performed without censoring at permanent discontinuation.
Time Frame: 12 months following acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE).
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Dabigatran Etexilate | Vitamin K Antagonist
Number analyzed (Participants) | 1681 | 1288
events per 100 patient-years | 1.61 [0.97 to 2.52] | 2.22 [1.38 to 3.40]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Vitamin K Antagonist; Test type: Other; p = 0.542, Regression, Cox — One-side p-value; Cox-regression proportional hazards model including fixed effects for treatment; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.299 to 1.885] — Hazard Ratio < 1 favors Dabigatran etexilate

8. Secondary Outcome: Objective 2: Incidence Rate of VTE-related Mortality
Description: Incidence rate of VTE-related Mortality per 100 patient-years (1/(100*patient-years)). Each patient in the two treatment groups was weighted proportionally to the probability of that patient being assigned to the opposite treatment group, conditional on relevant observed baseline variables. The propensity scores were estimated using the multivariable logistic regression model.
  For the restricted patient set, as a sensitivity analysis, the calculation of incidence rates and cumulative risks was performed without censoring at permanent discontinuation.
Time Frame: 12 months following acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE).
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Dabigatran Etexilate | Vitamin K Antagonist
Number analyzed (Participants) | 1681 | 1288
events per 100 patient-years | 0 [0 to 0] | 0.42 [0.11 to 1.08]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Vitamin K Antagonist; Test type: Other; p = 0.996, Regression, Cox — One-side p-value; Cox-regression proportional hazards model including fixed effects for treatment; Hazard Ratio (HR) = 0.00 — Hazard Ratio < 1 favors Dabigatran etexilate. Hazard Ratio is actually <0.01 95% Confidence Interval is not calculable (NA) due to insufficient number of participants with events

9. Secondary Outcome: Objective 2: Incidence Rate of All-cause Mortality
Description: Incidence rate of all-cause mortality per 100 patient-years (1/(100*patient-years)). Each patient in the two treatment groups was weighted proportionally to the probability of that patient being assigned to the opposite treatment group, conditional on relevant observed baseline variables. The propensity scores were estimated using the multivariable logistic regression model.
  For the restricted patient set, as a sensitivity analysis, the calculation of incidence rates and cumulative risks was performed without censoring at permanent discontinuation.
Time Frame: 12 months following acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE).
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Dabigatran Etexilate | Vitamin K Antagonist
Number analyzed (Participants) | 1681 | 1288
events per 100 patient-years | 2.12 [1.37 to 3.12] | 3.06 [2.05 to 4.39]
Statistical Analysis 1: Comparison: Dabigatran Etexilate vs Vitamin K Antagonist; Test type: Other; p = 0.690, Regression, Cox — One-side p-value; Cox-regression proportional hazards model including fixed effects for treatment; Hazard Ratio (HR) = 0.857, 95% CI 2-sided [0.402 to 1.828] — Hazard Ratio < 1 favors Dabigatran etexilate

ADVERSE EVENTS:
Time Frame: From the time of VTE until the end of the study (Dabigatran etexilate (1) and (2) and Vitamin K antagonist (1) and (2)) or from the time of informed consent until the end of the study (not assigned to Dabigatran etexilate or Vitamin K antagonist), up to 12 months.
Description: Adverse events are reported based on all eligible patients.
Arm/Group | Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist | Dabigatran Etexilate (1) | Dabigatran Etexilate (2) | Vitamin K Antagonist (1) | Vitamin K Antagonist (2)
All-Cause Mortality (participants affected / at risk) | 54/3714 | 13/1006 | 42/910 | 25/1375 | 30/792
Serious Adverse Events (participants affected / at risk) | 60/3714 | 22/1006 | 47/910 | 34/1375 | 41/792
Other Adverse Events (participants affected / at risk) | 0/3714 | 0/1006 | 0/910 | 0/1375 | 0/792
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Assigned to Dabigatran Etexilate or Vitamin K Antagonist (N=3714) | Dabigatran Etexilate (1) (N=1006) | Dabigatran Etexilate (2) (N=910) | Vitamin K Antagonist (1) (N=1375) | Vitamin K Antagonist (2) (N=792)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 5 | 0 | 5 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 4 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Right-to-left cardiac shunt (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 2
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 7 | 3 | 6 | 7 | 7
Drug intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 2
Sepsis (Infections and infestations) | 3 | 0 | 1 | 2 | 0
Septic shock (Infections and infestations) | 3 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 1 | 2
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebellar haematoma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Coma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 1 | 1 | 0
Nephroptosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Arterial rupture (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Internal haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT02596230/SAP_000.pdf
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT02596230/Prot_001.pdf